CLINICAL TRIAL: NCT01344941
Title: Human Immune Responses Toward HIV-1 Envelope Antigens
Acronym: HIVBLD
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XPD09-022 HIVBLD
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: HIV Infection
Keywords: Vaccine response; Human Lymphocytes
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maximally, there will be up to 30 draws per study participant with no more than 120 ml of blood collected at any one time and no more than 2.5 L collected for the entire study. Samples will be used for continued B-cell and T-cell studies supportive of the 2 study objectives. The volume of blood drawn will be closely monitored and will remain below the defined criteria for minimal risk research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: The first group will comprise individuals who have received a St. Jude HIV-1 vaccine and who have exhibited sustained immune responses
- Group 2: Groups 2 will be HIV-1-infected. The first visit of individuals in groups 2 will involve the collection of 120 ml of blood as well as a minimal blood volume required for the specified screening laboratory evaluation for each group.
- Group 3: Groups 3 will be HIV-1-uninfected. The first visit of individuals in groups 3 will involve the collection of 120 ml of blood as well as a minimal blood volume required for the specified screening laboratory evaluation for each group.

SUMMARY:
The primary objectives of this study is to

* Define the envelope-specific B-cell and T-cell responses in humans who have received a St. Jude HIV-1 vaccine.
* Describe mechanisms of HIV-1 envelope processing and consequent B-cell and T-cell activities.

DETAILED DESCRIPTION:
The goal of this protocol is to understand how human lymphocytes respond to HIV-1 antigens in the context of vaccination or infection. This protocol will support understanding of the immune response by providing a source of lymphocytes and serum from selected individuals to study in laboratory based investigations. Blood samples from individuals who have received an HIV-1 vaccine, individuals who are HIV-1-infected, and individuals who are HIV-1-uninfected are requested to: (1) test previously vaccinated volunteers for HIV-1 envelope-specific B-cell and T-cell immune activities, and (2) increase understanding of how the human immune system processes and responds to HIV-1 envelope proteins.

ELIGIBILITY:
Inclusion Criteria:

* Participant is greater than or equal to 18 years of age.
* Participant is in good general health.
* Participant weighs ≥ 110 pounds.
* Participant has hemoglobin > 12 gm/dL within last 12 weeks.

Group 1 (Vaccinees) only Inclusion Criteria:

* Participant has previously received one of the St. Jude HIV-1 vaccines via enrollment in prior St. Jude HIV vaccine studies.

Group 2 (HIV positive) only Inclusion Criteria:

* Participant is HIV-1 positive by medical record review.

Group 3 (HIV negative) only Inclusion Criteria:

* Participant is HIV-1 negative as determined by HIV ELISA.

Exclusion Criteria:

* Participant is unable or unwilling to give written informed consent.
* Participant is pregnant female.

Group 2 (HIV positive) only Exclusion Criteria:

* Participant is enrolled in other clinical trials that include any blood sampling such that the cumulative blood draws would exceed that established as constituting minimal risk (e.g., more than 550 ml in an 8 week period with collection more frequently than 2 times per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Previous St. Jude HIV-1 vaccine study participants will be contacted by phone by study investigators or their designees to assess interest in participation in this protocol.
  Group 2: Participants will be recruited from those receiving care for their HIV infection in the Translational Trials Unit at St. Jude.
  Group 3: Participants will be recruited from the Memphis community. Recruitment will occur on College and University campuses, from community groups, through word-of-mouth, and through the use of a study brochure.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Specific B cell and T cell responses in humans who received St Jude HIV-1 Vaccine | 5 years
  The outcome measures will be assessed in such a way that individuals will be sampled longitudinally (every 6months) until the immune response is no longer detectable by HIV ELISA or until the 5 year study period is complete, whichever comes first. A volume of 120 ml will be collected at each visit for immune response assays (both B-cell and T-cell) and 2 ml of blood will be collected for the HIV ELISA.

SECONDARY OUTCOMES:
Mechanism of HIV-1 envelope processing B cell and T cell activities | 5 years
  The outcome measures will be assessed by new developments in the field that may ultimately yield improved methods for the testing of antigen processing and B-cell and T-cell functions, in which case new assays will be adopted for use in this study. Lymphocyte samples will also support HLA testing. Samples will be used for continued B-cell and T-cell studies supportive of the 2 study objectives. The volume of blood drawn will be closely monitored and will remain below the defined criteria for minimal risk research.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Flynn, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols